CLINICAL TRIAL: NCT06573918
Title: EMG-Assessed Paratonia: A Novel Approach to Investigating Motor Response Inhibition in Healthy Subjects
Brief Title: EMG-Assessed Paratonia: A New Approach to Response Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Luca Puce, Principal investigatior, Universita degli Studi di Genova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EMG-DINOGMI-2024
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Electromyography Physical activity; Motor inhibition; Frontal circuits; Sport-specific

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMG-assessed paratonia group (Experimental): The study evaluated EMG-assessed paratonia to measure motor response efficiency across three groups of healthy young adults with varying physical activity levels: professional athletes (in both open and closed skills sports), amateurs, and sedentary individuals. Surface electrodes were placed on the biceps and triceps brachii muscles during passive elbow movements while participants remained relaxed. EMG activity detected during these movements was used to quantify the level of paratonia, indicating the participants' ability to relax their muscles.
  Interventions: Diagnostic Test: EMG-based assessment of paratonia

INTERVENTIONS:
Diagnostic Test: EMG-based assessment of paratonia — EMG-assessed paratonia was analyzed and compared to assess motor response efficiency in three groups of healthy young adults with different levels of physical activity: professional athletes engaged in closed and open skills sports, amateurs, and sedentary individuals. To analyze EMG-assessed paratonia, two surface electrodes were attached to the biceps and triceps brachii muscles during passive flexion-extension movements of the elbow while the participant remained in a state of maximum relaxation. Any EMG activity detected during these movements was attributed to an inability to relax, thereby reflecting their degree of paratonia.

SUMMARY:
Paratonia is the inability to relax muscles during the assessment of muscle tone in the absence of spasticity and parkinsonian rigidity. It can be evaluated qualitatively using clinical scales and objectively through surface electromyography (EMG-assessed paratonia). It is widely accepted that paratonia represents a manifestation of impaired motor response inhibition due to frontal lobe dysfunction.

Traditionally, motor response inhibition has been assessed using experimental protocols such as go/no-go and stop-signal tasks. Research has shown that athletes, particularly those engaged in open-skill sports, demonstrate superior motor response inhibition compared to sedentary individuals. Even amateur athletes exhibit better motor response inhibition than sedentary individuals, though to a lesser extent than professional athletes.

Given that the etiology of paratonia involves a defect in motor response inhibition, it is hypothesized that EMG-assessed paratonia could become a novel approach for evaluating motor response inhibition. The present study was designed to validate this hypothesis. Specifically, we first tested whether EMG-assessed paratonia in healthy subjects can reveal a well-known aspect of motor response inhibition, namely its correlation with the level of physical activity.

DETAILED DESCRIPTION:
EMG-assessed paratonia was analyzed and compared to assess motor response efficiency in three groups of healthy young adults with different levels of physical activity: professional athletes engaged in closed and open skills sports, amateurs, and sedentary individuals. To analyze EMG-assessed paratonia, two surface electrodes were attached to the biceps and triceps brachii muscles during passive flexion-extension movements of the elbow while the participant remained in a state of maximum relaxation. Any EMG activity detected during these movements was attributed to an inability to relax, thereby reflecting their degree of paratonia.

ELIGIBILITY:
Inclusion Criteria:

Sedentary Individuals: Defined as those engaging in less than 16.67 metabolic equivalent of task (MET) hours per week.

Amateur Athletes: Defined as individuals who engage in 16.67 to 25 MET hours per week.

Professional Athletes: Defined as individuals who engage in more than 25 MET hours per week.

Exclusion Criteria:

Presence of any pathology or pain in the flexor or extensor muscles of the arm. Use of muscle stimulants, relaxants, steroids, tobacco, alcohol, or any other drugs.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Neuromuscular excitation of the Biceps Brachii (paratonia assessed by EMG) during passive elbow flexion and extension | Throughout the duration of the evaluation, which lasts about 120 seconds
  Amplitude of electromyography value (Root Mean Square in microvolt) measured for Biceps Brachii muscle
Neuromuscular excitation of the Triceps Brachii (paratonia assessed by EMG) during passive elbow flexion and extension | Throughout the duration of the evaluation, which lasts about 120 seconds
  Amplitude of electromyography value (Root Mean Square in microvolt) measured for Triceps Brachii muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Genova, Genova, Italy